CLINICAL TRIAL: NCT01611766
Title: Evaluation of Secondary Cytoreductive Surgery in Platinum-Sensitive Recurrent Ovarian Cancer: A Phase III, Multicenter, Randomized Trial
Brief Title: Surgery or Chemotherapy in Recurrent Ovarian Cancer (SOC 1 Trial)?
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Gynecologic Oncology Group (Other Government)
Collaborators: Fudan University (Other); Zhejiang Cancer Hospital (Other); Shanghai Zhongshan Hospital (Other); Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGOG OV 2; SGOG OV2 (Other: SGOG)
Record Dates: First submitted 2012-05-30; First posted 2012-06-05 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Ovarian Epithelial Cancer Recurrent; Fallopian Tube Carcinoma; Primary Peritoneal Carcinoma
Keywords: secondary cytoreductive surgery; Ovarian Cancer; surgery; recurrence
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- secondary cytoreductive surgery (Experimental): SCR followed by chemotherapy
  Interventions: Procedure: Secondary Cytoreductive Surgery; Drug: Salvage Chemotherapy
- Salvage Chemotherapy (Active Comparator): platinum-based chemotherapy
  Interventions: Drug: Salvage Chemotherapy

INTERVENTIONS:
Procedure: Secondary Cytoreductive Surgery — Complete Cytoreduction
  Other Names: Maximum effort cytoreductive surgery
  Arms: secondary cytoreductive surgery
Drug: Salvage Chemotherapy — 6 cycles of postoperative chemotherapy
  Other Names: second line chemotherapy

SUMMARY:
The purpose of this study is to evaluate the role of secondary cytoreduction (SCR) and validate the risk model of patient selection criteria in platinum-sensitive recurrent ovarian cancer.

DETAILED DESCRIPTION:
The primary objective is to determine whether secondary cytoreduction followed by chemotherapy is superior to chemotherapy alone in improving progression-free survival (PFS) and overall survival (OS) in patients with platinum-sensitive recurrent ovarian cancer

ELIGIBILITY:
Inclusion Criteria:

* Age at recurrence ≥ 18 years
* Patients with platinum-sensitive, first relapsed epithelial ovarian, primary peritoneal, or fallopian tube cancer (EOC, PPC, FTC), which is defined as those with treatment -free interval of 6 months or more.
* A complete secondary cytoreduction predicting score, iMODEL [Tian WJ, Ann Surg Oncol 2012,19(2):597-604]<=4.7, including FIGO stage (0 or 0.8); residual disease after primary surgery (0 or 1.5); Progression-free interval (0 or 2.4); PS ECOG (0 or 2.4); Ca125 (0 or 1.8); and ascites at recurrence (0 or 3.0). If PI and CO-PI reach consensus that the recurrent tumor detected by PET/CT could be completely resected, the index of CA125 could be scored as 0. (Revised on 09/30/2013)
* Assessed by the experienced surgeons, complete resection of all recurrent disease is possible. If single lesion outside the peritoneal cavity can be resected, MRI/CT or PET/CT scan should be performed to exclude simultaneous intra-abdominal lesions.
* Patients who have given their signed and written informed consent and their consent.

Exclusion Criteria:

* Patients with borderline tumors as well as non-epithelial tumors.
* Patients for interval-debulking, or for second-look surgery, or palliative surgery planned.
* Impossible to assess the resectability or evaluate the score. Radiological signs suggesting complete resection is impossible.
* More than one prior chemotherapy.
* Second relapse or more
* Patients with second or other malignancies who have been treated by surgery, if the treatment might interfere with the treatment of relapsed ovarian cancer or if major impact on prognosis is expected.
* Progression during chemotherapy or recurrence within 6 months after first-line therapy
* Any contradiction not allowing surgery and/or chemotherapy

  1. Accompanied by hypoxia serious chronic obstructive pulmonary disease
  2. Uncontrolled hypertension, cerebrovascular accident/ Stroke, myocardial infarct, unstable angina, untreated thrombosis, chronic congestive heart failure, or serious arrhythmia in need of medicine.
  3. Severe hepatitis, history of liver disease, nephrotic syndrome, renal insufficiency
  4. Active ulcer history, abdominal wall fistula, perforation of gastrointestinal tract, or Intra-abdominal abscess, or simultaneously apply treatment/prevent ulcers therapy.
  5. Uncontrolled diabetes
  6. Uncontrolled epilepsy need long-term antiepileptic treatment.
* Any medication induced considerable risk of surgery, e.g. estimated bleeding due to oral anticoagulating agents, or bevacizumab.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2012-07-19 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Up to 60 months after last patient randomized
  from date of randomisation until death
Progression-free survival | Up to 24 months after last patient randomized
  interval between date of randomization and the date of second relapse/ progression or death, whatever occurs first

SECONDARY OUTCOMES:
Accumulating Treatment-free survival (TFSa) | Up to 60 months after last patient randomized
  the time of OS minus each treatment period after randomization, including surgery and chemotherapy
Overall survival after the adjustment of one-way treatment switching | Up to 60 months after last patient randomized
  OS adjusted by statistical models for crossover
30-day post-operative complications | From the operation until after 30 days
  MSKCC surgical complications grading method and CTCAE v4.03 criteria will be adopted for evaluating the perioperative complications
Validation of iMODEL | From randomization to operation
  iMODEL score to predict complete resection
Patient compliance | Up to 60 months after last patient randomized
  compliance with protocol
Quality of life assessments | Study entry; 6 months; 12 months; 24 months and 60 months after randomization
  The EORTC core quality of life questionnaire (QLQ-C30, version 3.0) Functional Assessment of Cancer Therapy- Ovary (FACT-O)
Time to first subsequent anticancer therapy | Up to 60 months after last patient randomized
  From date of randomization until the date of first recurrent anticancer therapy
Time to second subsequent anticancer therapy | Up to 60 months after last patient randomized
  From date of randomization until the date of secondary recurrent anticancer therapy

CONTACTS AND LOCATIONS:
Overall Officials: Rongyu Zang, MD,PhD, Principal Investigator — Shanghai Gynecologic Oncology Group
Locations (4):
- China (4):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Fudan University Cancer Hospital, Shanghai, Shanghai Municipality
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Jiang R, Feng Y, Chen Y, Cheng X, Shi T, Gao W, Jia H, Jiang S, Guo Y, Huang X, Tu D, Zhang Y, Yang H, Zhang P, Liu J, Zhu J, Zang R; SOC-1 Investigators. Surgery versus no surgery in platinum-sensitive relapsed ovarian cancer: final overall survival analysis of the SOC-1 randomized phase 3 trial. Nat Med. 2024 Aug;30(8):2181-2188. doi: 10.1038/s41591-024-02981-0. Epub 2024 Jun 1. PMID 38824243
- [Derived] Shi T, Zhu J, Feng Y, Tu D, Zhang Y, Zhang P, Jia H, Huang X, Cai Y, Yin S, Jiang R, Tian W, Gao W, Liu J, Yang H, Cheng X, Zang R. Secondary cytoreduction followed by chemotherapy versus chemotherapy alone in platinum-sensitive relapsed ovarian cancer (SOC-1): a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2021 Apr;22(4):439-449. doi: 10.1016/S1470-2045(21)00006-1. Epub 2021 Mar 8. PMID 33705695
- See also: Shanghai Gynecologic Oncology Group — http://www.ShanghaiGOG.org